CLINICAL TRIAL: NCT05552937
Title: A Phase II, Single-Arm, Open-Label, Multicentre Study to Evaluate the Safety and Efficacy of Tafasitamab Combined With Lenalidomide in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Brief Title: Evaluate the Safety and Efficacy of Tafasitamab Combined With Lenalidomide in Patients With Relapsed or Refractory DLBCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-00901
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: DLBCL
MeSH Terms: interventions — tafasitamab; Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tafasitamab and Lenalidomide (Experimental): Tafasitamab and lenalidomide will be coadministered for up to 12 cycles (28 days per cycle).followed by tafasitamab monotherapy (in participants with stable disease or better) until treatment withdrawal criteria are met.
  Interventions: Drug: Tafasitamab and Lenalidomide

INTERVENTIONS:
Drug: Tafasitamab and Lenalidomide — Tafasitamab will be administered intravenously in 28-day cycles. During Cycles 1 through 3, tafasitamab will be administered weekly on Days 1, 8, 15, and 22; an additional loading dose will be administered on Cycle 1 Day 4. Starting with Cycle 4, tafasitamab will be administered on Days 1 and 15 of each cycle.
  Participants will self-administer lenalidomide capsules orally on Days 1-21 of each 28-day cycle, up to 12 cycles.

SUMMARY:
This is a A Phase II, Single-Arm, Open-Label, Multicentre Study to Evaluate the Safety and Efficacy of Tafasitamab Combined with Lenalidomide in Patients with Relapsed or Refractory Diffuse Large B-Cell Lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years.
2. Histologically confirmed diagnosis of DLBCL not otherwise specified (NOS); T cell/histiocyte rich large B-cell lymphoma (THRLBCL); Epstein-Barr virus (EBV) positive DLBCL of the elderly (EBV-positive DLBCL), Grade 3b Follicular Lymphoma, Composite lymphoma with a DLBCL component with a subsequent DLBCL relapse, according to the Revised European American Lymphoma/World Health Organization (REAL/WHO) classification. Additionally, patients with the evidence of histological transformation to DLBCL from an earlier diagnosis of low grade lymphoma (i.e., an indolent pathology such as follicular lymphoma, marginal zone lymphoma, chronic lymphocytic leukaemia) into DLBCL with a subsequent DLBCL relapse are also eligible.
3. Patients received at least one, but no more than three previous systemic regimens for the treatment of DLBCL and one therapy line must have included a CD20-targeted therapy.
4. Patients must meet the following laboratory criteria at screening.
5. Patients must use an effective barrier method of contraception.
6. In the opinion of the investigator the patients must be able and willing to receive adequate prophylaxis and/or therapy for thromboembolic events; be able to understand the reason for complying with the special conditions of the pregnancy prevention risk management plan and give written acknowledgement of this.

Exclusion Criteria:

1. Patients who have other histological type of lymphoma，primary refractory DLBCL，a history of "double/triple hit" genetics.
2. Patients who have, within 14 days prior to Day 1 dosing:

   1. not discontinued CD20-targeted therapy, chemotherapy, radiotherapy, investigational anticancer therapy or other lymphoma specific therapy.
   2. undergone major surgery or suffered from significant traumatic injury.
   3. received live vaccines.
   4. required parenteral antimicrobial therapy for active, intercurrent infections.
3. Patients who:

   1. were previously treated with CD19-targeted therapy or IMiDs® (e.g. thalidomide, LEN).
   2. have undergone ASCT within the period ≤ 3 months prior to signing the informed consent form.
   3. have undergone previous allogenic stem cell transplantation.
   4. have a history of deep venous thrombosis/embolism and who are not willing/able to take venous thromboembolic event prophylaxis during the entire treatment period.
   5. concurrently use other anticancer or experimental treatments.
4. Prior history of malignancies other than DLBCL.
5. Patients with:

   1. positive hepatitis B and/or C serology.
   2. known seropositivity for or history of active viral infection with human immunodeficiency virus (HIV).
   3. CNS lymphoma involvement.
   4. history or evidence of clinically significant cardiovascular, CNS and/or other systemic disease that would in the investigator's opinion preclude participation in the study or compromise the patient's ability to give informed consent.
   5. history or evidence of severe hepatic impairment (total serum bilirubin > 3 mg/dL).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 1-3 years approximately
  Evaluation by the Independent Review Committee (IRC).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 1-3 years approximately
  Evaluated by the IRC according to cheson 2007 and cheson 2014.
Disease Control Rate (DCR) | 1-3 years approximately
Duration of Response (DOR) | 1-3 years approximately
Progression Free Survial (PFS) | 1-3 years approximately
Time to progression (TTP) | 1-3 years approximately
Time to response (TTR) | 1-3 years approximately
Overall Survival (OS) | 1-3 years approximately
Safety of Lenalidomide combined with Tafasitamab according to the frequency and severity of adverse events (AEs). | 2 years
Potential immunogenicity of Tafasitamab. | 2 years
Maximum serum concentration (Cmax) | 2 years
Time to maximum serum concentration (tmax) | 2 years
Apparent trough serum concentration before dosing (Cpd) | 2 years
Area under the serum concentration versus time curve from time 0 to the time t of the last quantifiable concentration (AUC0-t) | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The First Afflicated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] You J, Chen W, Yan Z, Tian D, Yi H, Feng Y, Zhang M, Xing T, Wang Z, Zhao W, Xu P. Anti-CD19 antibody tafasitamab therapy for relapsed or refractory diffuse large B-cell lymphoma: a case series. Anticancer Drugs. 2026 Feb 1;37(2):123-127. doi: 10.1097/CAD.0000000000001774. Epub 2025 Oct 30. PMID 41176775